CLINICAL TRIAL: NCT04094220
Title: A Randomized, Controlled Trial of Lateral Lumbar Interbody Fusion Plus Posterior Decompression or Not for Severe Lumbar Spinal Stenosis
Brief Title: LLIF Plus Posterior Decompression for Severe Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-161
Record Dates: First submitted 2019-08-26; First posted 2019-09-18 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2020-12

CONDITIONS: Lumbar Spine Degeneration; Lumbar Spinal Stenosis
Keywords: indirect decompression; lateral interbody fusion; lumbar; direct decompression
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Patients included in this study are with degenerative lumbar stenosis and Schizas's stenosis grades C. Patients who suffered from significant lumbar scoliosis, grade 2 spondylolisthesis, lumbar fracture and prior lumbar surgery are excluded from this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral lumbar interbody fusion (Experimental): Patients in this group received lateral lumbar interbody fusion alone. Patients who suffered residual neurologic symptoms postoperatively will received conservative treatment for at least 3 months.Patients were considered to have unsuccessful indirect decompression if they had less than 20% improvement according to the Oswestry Disability Index (ODI) by 3 months postoperatively.
  Interventions: Procedure: Lateral lumbar interbody fusion
- Lateral lumbar interbody fusion plus posterior decompression (Experimental): Patients in this group received lateral lumbar interbody fusion plus posterior decompression.
  Interventions: Procedure: Lateral lumbar interbody fusion

INTERVENTIONS:
Procedure: Lateral lumbar interbody fusion — LLIF is an indirect decompression technique, and does not directly remove the disc or osteophyte protruding into the spinal canal. Its decompression effect is not as thorough as traditional posterior decompression surgery. Usually, posterior decompression is required for patients who have unsuccessful indirect decompression.

SUMMARY:
Lateral lumbar interbody fusion (LLIF), as a minimally invasive technique, is an indirect decompression technique, and its decompression effect is not as thorough as traditional posterior decompression surgery. For certain patients with severe lumbar stenosis, additional posterior decompression is required. However, whether additional posterior decompression is necessary for these patients is unknown. Radiographic predictors of failed indirect decompression via LLIF is unknown. In current randomized, controlled trial , the investigators compare the clinical outcomes of patients with severe lumbar stenosis who received LLIF plus posterior decompression and those without posterior decompression.

DETAILED DESCRIPTION:
The current randomized controlled trial consists of two groups. Patients included in the study are with Schizas's stenosis grades C. Patients in one group received transpsoas lateral lumbar interbody fusion. Patients in the other group received transpsoas lateral lumbar interbody fusion plus posterior decompression. Patients will be followed for one year. Clinical outcomes of the two groups will be compared. And radiographic predictors of failed indirect decompression via LLIF will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who are 50 - 80 years of age.
* Patients who present with symptomatic Grade I or II degenerative spondylolisthesis at one or two contiguous lumbar levels between L1 and L5 and who are surgical candidates for interbody lumbar fusion surgery; symptoms should include radiculopathy and/or neurogenic claudication with or without back pain.
* Patients who have been unresponsive to at least 6 months of conservative treatments or who exhibit progressive neurological symptoms in the face of conservative treatment.
* Patients who understand the conditions of enrollment and are willing to sign an informed consent to participate in the study.

Exclusion Criteria:

* Patients with lumbar pathologies requiring treatment at more than two levels.
* Patients who have had previous lumbar fusion surgery.
* Patients with congenital lumbar stenosis.
* Patients with radiographic confirmation of Grade IV facet joint disease or degeneration.
* Patients with noncontained or extruded herniated nucleus pulposus.
* Patients with active local or systemic infection.
* Patients with rheumatoid arthritis or other autoimmune disease.
* Patients who cannot undergo magnetic resonance imaging (MRI).
* Patients who are mentally incompetent.
* Patients with BMI over 30kg/m2 or less than 18 kg/m2.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Preoperative, 3-month, 12-month,24-month after surgery
  The ODI is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Preoperative, 3-month, 12-month,24-month after surgery
  The VAS is a self-report measure of the intensity of pain (score range 0 - 10 ). A higher score indicates greater pain intensity.
Zurich Claudication Questionnaire(ZCQ) | Preoperative, 3-month, 12-month,24-month after surgery
  The ZCQ is a disease-specific self-report outcome instrument commonly used in trials to measure treatment outcomes in patients with lumbar spinal stenosis.The result is expressed as a percentage of the maximum possible score (22.22% - 100%). The score increases with worsening disability.The The ZCQ consists of three subscales: symptom severity scale, physical function scale and patient's satisfaction with treatment scale.

OTHER OUTCOMES:
Axial central canal area | Preoperative,postoperative,12-month,24-month after surgery
  The area of the spinal central canal with the most stenosis at the level of the intervertebral disc on MRI.
Midsagittal canal diameter | Preoperative,postoperative,12-month,24-month after surgery
  The canal diameter at the midsagittal slice on MRI.
anterior and posterior disc height | Preoperative,postoperative, 6-month,12-month,24-month after surgery
  The disc height at the anterior and posterior rim of the intervertebral disc on X-ray.
The height of the bilateral intervertebral foramen | Preoperative,postoperative, 6-month,12-month,24-month after surgery
  The distance of minimum diameter between adjacent pedicles on CT.
Disc angle | Preoperative,postoperative, 6-month,12-month,24-month after surgery
  The angles of the lines parallel to the upper and lower endplates in the intervertebral space.

CONTACTS AND LOCATIONS:
Overall Officials: Fangcai Li, MD, Principal Investigator — The Second Affiliated Hospital of Medical College Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Medical College Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No